CLINICAL TRIAL: NCT07336017
Title: Impact on Postpartum Anal Incontinence of an Educational Program for Delivery Room Staff on the Diagnosis and Repair of Obstetric Anal Sphincter Injuries
Brief Title: Impact on Postpartum Anal Incontinence of an Educational Program for Delivery Room Staff
Acronym: IIA-LOSA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9694
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Anal Incontinence
Keywords: Anal Incontinence; Postpartum Anal Incontinence; Obstetric Anal Sphincter Injuries
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstetric anal sphincter injuries are a source of significant short-term (pain, bleeding, infection, suture dehiscence), medium-term (anorectovaginal fistulas, sexual dysfunction), and long-term (anal incontinence in 30-60% of cases) morbidity. However, they are underdiagnosed and sometimes poorly repaired due to technical difficulties, the use of inappropriate surgical techniques, or a lack of awareness of their significant long-term morbidity. These diagnostic and therapeutic errors, however, significantly worsen the functional prognosis of patients. This study aims to evaluate the clinical impact of an educational program designed for continuing education in the diagnosis and repair of obstetric anal sphincter injuries for staff working in the delivery room.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (≥18 years old)
* who gave birth vaginally at Strasbourg University Hospital in the 3 months prior to and 3 months following the training of delivery room staff at both maternity wards
* Singleton pregnancy
* Live birth

Exclusion Criteria:

* Multiple pregnancy
* Fetal death in utero
* Medical termination of pregnancy
* Delivery by cesarean section.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women (≥18 years old) who gave birth vaginally at Strasbourg University Hospital in the 3 months prior to and 3 months following the training of delivery room staff at both maternity wards
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
St. Mark's score | Up to 18 months
  The St Mark's score is a tool for measuring the severity of fecal incontinence:
  The score is based on several criteria:
  Solid leakage: 2 points (1-3 times per month) Liquid leakage: 3 points (once a week) Gas: 1 point (less than once a week) Protection: 1 point (occasionally) Daily life: 2 points (moderate discomfort) Ability to control: 1 point
  The points for each criterion are added together:
  * Minimum score = 0 → no incontinence.
  * Maximum score = 24 → very severe incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologique et d'Obstétrique - CHU de Strasbourg - France, Strasbourg, France